CLINICAL TRIAL: NCT00184223
Title: Motivational Interviewing to Acutely Admitted Psychiatric Patients With Comorbid Substance Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GB-MI-2004
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-05

CONDITIONS: Substance-Related Disorders
Keywords: Motivational Interviewing; Substance abuse; Acuteley admitted psychiatric patients; Emergency Services, Psychiatric
MeSH Terms: conditions — Substance-Related Disorders | interventions — Motivational Interviewing; Therapeutics

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- motivational interviewing (Experimental): Manual guided motivational interviewing in addition to treatment as usual
  Interventions: Behavioral: Motivational Interviewing; Other: Treatment as usual
- control group (Other): treatment as usual
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Motivational Interviewing — 2 sessions of 45 minutes each with manual guided motivational interviewing delivered individually by a trained therapist.
  Arms: motivational interviewing
Other: Treatment as usual — Treatment as usual is individualized according to the clinical condition of the patients during the stay and in accordance with general national and international medical standards. It includes detoxification, pharmacotherapy, and general psychotherapy. Also, treatment is given for any coexisting non-substance-related disorder, including psychiatric disorders.

SUMMARY:
The purpose for this study is to determine whether 2x45 minutes Motivational Interviewing given during hospital stay to acutely admitted psychiatric patients with substance use problems, can reduce substance use after discharge.

DETAILED DESCRIPTION:
The aims of the study are in a randomized controlled trial to compare the effects of 2 x 45 minutes Motivational Interviewing and standard treatment with standard treatment alone.All patients acutely admitted to Østmarka Psychiatric Hospital are evaluated for substance use, and all patients with substance use that give their consent to participate are randomized to Motivational Interviewing and standard treatment or standard treatment alone.

Substance use and function will be followed for two years.Admittances to hospital and contacts with primary health care for five years.

ELIGIBILITY:
Inclusion Criteria:

* substance use
* acutely admitted to psychiatric hospital

Exclusion Criteria:

* dementia
* serious brain damage
* not speaking Norwegian or English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2004-10; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Substance use and function questionnaire | 2 years

SECONDARY OUTCOMES:
Admissions to hospital | 2 years
Number of contacts with primary ealth care | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Morken, MD PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Østmarka Psychiatric Department, St. Olavs Hospital, University Hospital of Trondheim, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bagoien G, Bjorngaard JH, Ostensen C, Reitan SK, Romundstad P, Morken G. The effects of motivational interviewing on patients with comorbid substance use admitted to a psychiatric emergency unit - a randomised controlled trial with two year follow-up. BMC Psychiatry. 2013 Mar 21;13:93. doi: 10.1186/1471-244X-13-93. PMID 23517244